CLINICAL TRIAL: NCT01394471
Title: Oxytocin Treatment of Social Cognitive and Functional Deficits in Schizophrenia
Acronym: OTS-12WK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cort Pedersen, MD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0259; R01MH093529 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; oxytocin; OT; social cognition; social functioning; paranoia; psychosis; psychotic symptoms; social deficits; intranasal administration
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Social Adjustment; Paranoid Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxytocin (Experimental): Twice daily treatment of oxytocin will be administered by subjects
  Interventions: Drug: Intranasal Oxytocin Spray
- Control spray (Placebo Comparator): Self administration twice daily of intranasal spray that does not contain oxytocin
  Interventions: Drug: Intranasal Oxytocin Spray

INTERVENTIONS:
Drug: Intranasal Oxytocin Spray — 6 insufflations (24IU of oxytocin total) given twice daily for 12 weeks
  Other Names: Syntocinon spray

SUMMARY:
Purpose: Test whether intranasal administration of the neuropeptide, oxytocin, improves social cognition, psychotic symptoms and social functioning in schizophrenia.

Participants: 80 adults with schizophrenia or schizoaffective disorder for at least one year.

Procedures (methods): Oxytocin or placebo will be administered twice daily in an intranasal spray for 12 weeks. Before, during and at the end of the trial, each subject will undergo psychiatric symptom ratings and tests of mental abilities used in social functioning, cognition, and social competence.

DETAILED DESCRIPTION:
Overview of Procedures: All procedures will be conducted at the UNC Hospitals Clinical and Translational Research Center (CTRC) outpatient clinic or at the outpatient North Carolina Psychiatric Research Center (NCPRC), a specialized program of the University of North Carolina Center for Excellence in Community Mental Health in Raleigh, NC. Except for Screening, all clinic visits will begin between 0800-1000 hours and subjects will have fasted since midnight. Approximately 10 minutes after checking into the clinic, subjects' weight and vital signs will be measured followed by blood and urine sample collection. Breakfast will then be served. At regular intervals during each clinic visit, subjects will be allowed to rest for 15-20 minutes. Lunch will also be provided for the subjects.

Screening assessment: During the initial clinic visit and after giving informed consent, prospective subjects' psychiatric and medical histories will be reviewed, physical exams conducted, EKGs run and blood and urine collected for complete blood count (CBC), electrolytes, liver/renal function tests, TSH, glucose, urinalysis (UA), pregnancy test, and urine drug screen (UDS). The Structured Clinical Interview for DSM-IV will be administered to confirm diagnoses if one not on record within the past two years. The WRAT will be administered to determine reading ability as well as the Reading the Mind in the Eyes Test (Eyes Test) to determine if subjects meet the social cognition criterion for impairment. Finally, PANSS and Calgary Depression Scale ratings will be obtained.

Baseline and Treatment Week 6 and 12 assessments: All of the primary and secondary outcome measures will be obtained during clinic visits at Baseline (occurring within 1 week after the Screening assessment) and at the end of the treatment trial (12-week time point). Some of the outcome measures will be obtained at a clinic visit at the 6-week time point during the treatment trial. Subjects will arrive at the clinic between 8:00 and 10:00 a.m. for each of these visits where they will be given breakfast. At Baseline, administration of assessments will begin 10 min after completion of breakfast. At the 6 and 12-week clinic visits, assessments will begin 50 min after intranasal administration of test treatment (which will be given before breakfast-see details below). The primary outcomes are social cognition measures (details below): emotion recognition (ER-40, Eyes Test), theory of mind (Eyes Test, Brüne test), social perception (Trustworthiness Task) and attributional style (AIHQ). The secondary outcomes (details below) are social functioning (SLOF), social skill (role plays), psychotic symptoms (PANSS), paranoia (Green Paranoia Thought Scale), empathy (IRI), non-social cognition (RBANS), anxiety (Liebowitz social anxiety scale) depression (Calgary Depression Rating Scale), social perception (IPT-15) and food cravings (Food Craving Inventory and Night Eating Questionnaire). While we ultimately want to improve social functioning, we acknowledge that this domain might be slower to improve than social cognition, thus rendering it a secondary rather than primary outcome (and for that reason, we are assessing social functioning only at baseline and week 12 (end of treatment)). We included non-social cognition in the battery to assess whether treatment effects on social cognition generalize to other domains of cognition. A similar sentiment underlies our inclusion of symptoms (both psychotic and general) in the battery, as the value of OT may be enhanced if it can impact symptoms that might ultimately interfere with treatment engagement. Finally, we included empathy because of the relationship with theory of mind.

Test substance administration and other procedures during the treatment trial: During the treatment trial, subjects will self-administer test treatments twice daily; before breakfast and before dinner. Each treatment consists of 6 insufflations (each 0.1 ml) of Syntocinon Spray (Novartis), which contains 24 international units of OT, or placebo solution containing all of the ingredients in Syntocinon Spray except OT. Blind-labeled test treatment vials will be dispensed following a randomization scheme permuted in blocks of 4, stratified by gender, as oxytocin often has different effects in males and females, in animals and in humans. Subjects will self administer test treatments from 60 ml spray vials (ejecting 0.1 ml per spray) initially containing 35 ml of test substance. Each vial contains enough solution for 3 weeks of self administration. Subjects will receive their first vial of test treatment right after assessments are complete at the Baseline clinic visit. They will be instructed in intranasal self administration and care of test vials at that time and given written instructions on these matters. They will take their first intranasal test dose under the observation of research nurses before leaving the clinic. Before leaving the clinic, subjects will be given a card with the date of their return appointment in one week.

Subjects will return to the clinic at the 2, 6, 9 and 12 week time points during the treatment period. At the 2, and 9-week visits, subjects will have a brief visit with a study clinician who will assess side effects, perform a mental status examination, administer the PANSS and CGI. Spot urine pregnancy tests will also be done at the 2 and 9 week visits. At the baseline, 6 and 12-wk time points, subjects will arrive at the clinic between 8:00 and 10:00 a.m., having fasted overnight. Before eating breakfast, weight and vital sign measurements will be obtained along with blood and urine samples. Blood collected at baseline will be used to measure serum glucose and lipids and urine will be used to screen for pregnancy in women and for drug screening in all subjects. Blood and urine samples obtained at the 6 and 12-week time points will be used for the same measures obtained at the Screening visit. EKG will also be repeated at the 6 and 12-week time points. Prior to breakfast at the 6 and 12-wk time point visits, subjects will self-administer their morning dose while observed by a research nurse to be sure the process is being done correctly. To obtain plasma for later assay of OT concentrations, blood will be drawn 40 minutes after the morning test dose into a chilled EDTA vacutainer tube which will be immediately placed in an ice bath and spun down within 20 minutes. Plasma samples will be stored at ultralow temperatures. OT levels may reflect individual variability in OT absorption and metabolism and will be a covariate in statistical analyses.

Beginning 50 minutes after the morning test dose (6 and 12-week treatment time points), primary and secondary measures will be re-administered.

Subjects will bring their used test treatment vial to the clinic visits at the 2, 6, 9 and 12-week time points during the treatment trial. At the 2, 6 and 9 wk time points, subjects will be given a fresh test treatment intranasal spray vial from which they will continue twice daily self administration until the next visit. Subjects may be given two vials at the two week visit to ensure they have enough study medication until their week 6 visit.

Subjects will be called for two days following the baseline visit to remind them to take their study medication. They will then be called weekly for reminders for the remainder of the study (combined with check in call).

Randomization plan: The statistician (Dr. Hamer) will generate a randomization plan for randomizing 27 subjects to OT treatment and 27 subjects to placebo treatment using PROC PLAN in SAS Version 9.2. We will use a blocksize of 4 within each sex so that every 4 subject's randomization to the two groups will be equalized. The statistician will then export the randomization plan to a spreadsheet, which the data manager will import as a table into the study data management system.

When a subject is to be randomized, an authorized investigator (the data management systems we design allow different levels of functioning for each investigator) who does not need to be blinded will obtain the randomization number from the data management system. This authorized investigator will then contact the investigational drug service to give them the randomization number, and collect the appropriate medication from the investigational drug service.

Sources of test treatments: Dr. Pedersen has an IND exemption (#77,774) from the FDA to treat patients with schizophrenia with intranasal OT spray obtained from overseas pharmacies. The IND exemption is necessary because intranasal OT spray (Syntocinon Spray) has not been marketed in the USA since 1997 when Novartis let FDA approval of the product lapse for financial reasons (the product was not being prescribed frequently enough in this country to warrant the cost of maintaining FDA approval). Syntocinon Spray vials (5 ml) are ordered as needed from an international pharmacy. Triangle Compounding Pharmacy (Cary, NC) prepares each intranasal spray vial containing 35 ml of OT solution by decanting seven 5 ml Syntocinon Spray vials into a 60 ml spray vial. Triangle Compounding also prepares identical 60 ml spray vials containing 35 ml of a placebo solution that contains the same ingredients as Syntocinon Spray except for OT. OT in Syntocinon Spray remains stable for at least 1 month at room temperature.

Monitoring and enhancing compliance: Change in 60 ml spray vial weight over each 3-4 weeks of test treatment will be used to monitor subject compliance. Each insufflation (0.1 ml) should decrease the vial weight by 0.1 gram. Subjects will be called each week day morning to remind them to take their intranasal test treatment. Less than 75% of the anticipated decline in vial weight may be grounds for termination from the study, especially if it occurs more than once.

Monitoring safety: Laboratory tests, EKGs and vital signs will be obtained at the 6 and 12-week time points. Abnormalities or adverse events may result in exclusion from further participation. The Barnes, Simpson-Angus, and AIMS scales as well as a general side effects checklist will assist in thorough assessment of side effects.

Medical evaluation Screening: During the initial clinic visit and after giving informed consent, prospective subjects' psychiatric and medical histories will be reviewed, physical exams conducted, EKGs run and blood and urine collected for CBC, electrolytes, liver/renal function tests, TSH, glucose, UA, pregnancy test, and drug screen.

At baseline and during the treatment trial: An extensive set of lab values, EKGs and vital signs will be obtained during clinic visits at 6 and 12 weeks during the test treatment period (serum glucose and lipid measures will also be obtained at baseline). Subjects will have been fasting since midnight and will have not yet taken their morning test dose when their blood is drawn and urine collected shortly after they arrive for the baseline, week-6 and week-12 clinic visits. Running laboratory tests on blood and urine samples obtained in the fasting state, at these time points, is optimal for rapid detection of negative effects of OT treatment on subjects' physiology. It may also provide preliminary information about the influence of OT on the adverse metabolic effects of the atypical antipsychotic medications that most subjects will be taking throughout the study period. Vital signs will be repeated 2 hours after subjects take their morning intranasal test dose at the 6 and 12-week time points. Spot urine pregnancy tests will be obtained at screening, baseline, and weeks 2, 6, 9 and 12 clinic visits during the treatment trial.

Social Cognition Measures (Primary outcomes) The Emotion Recognition-40 Task (ER-40, Kohler et al 2004) consists of 40 faces presented sequentially on a computer screen along with the choices of rating the face as happy, sad, anger, fear or no emotion. It uses racially and ethnically diverse face images and is a psychometrically sound measure of social cognition in this clinical population (Carter et al 2009).

The Brüne Theory of Mind Stories Task (Brüne 2003) involves a series of 6 sets of 4 cartoon pictures that illustrate interactions between two or more individuals. The subject is asked to rearrange the pictures, initially presented in an illogical sequence, in an order that conveys a logical story. The period of time the subject takes to complete the task and the accuracy of the sequencing is recorded. Then, after the subject correctly organizes the pictures (which is done by the examiner if the subject's response is incorrect), the subject is asked questions about the cartoon characters' own beliefs and beliefs of other characters in the cartoons. The subject's interpretations of the characters' beliefs are scored as correct or incorrect.

The Reading the Mind in the Eyes test (Eyes Test, Baron-Cohen et al 2001) consists of 36 photographs and participants are asked to guess the mental state (i.e. what the person is thinking or feeling) from among 4 choice words. Participants are given a practice item to ensure that they understand the task. Each eye region is presented on a note card or is displayed on a computer screen with the four choice mental states shown in the four corners of the card or computer screen (one target word and three foil words). There is no time constraint in choosing the mental state. A glossary of the mental states is made available if the participants are unsure of the meaning of a word. Performance is measured by the number of faces correctly discriminated.

The Trustworthiness Task (Adolphs et al 1998) is comprised of 42 faces of unfamiliar people. Participants will be shown each picture individually (on a computer monitor) and will be asked to rate how much they would trust that person (i.e., with their money or their life) on a 7-point scale, ranging from -3 (very untrustworthy) to +3 (very trustworthy).

The Ambiguous Intentions Hostility Questionnaire (AIHQ, Combs et al 2007) is comprised of 15 short vignettes that reflect negative events that vary in intentionality (i.e., obvious, accidental, and ambiguous intentions). Participants are asked to read each vignette, to imagine the scenario happening to her/him (e.g., "You walk past a bunch of teenagers at a mall and you hear them start to laugh"), and to write down the reason why the other person (or persons) acted that way toward her/him (as a means of measuring attributions). Two independent raters subsequently code this written response for the purpose of computing a "hostility bias". The participant then rates, on Likert scales, whether the other person (or persons) performed the action on purpose (anchored by [1], definitely no, and [6], definitely yes), how angry it would make her/him feel (anchored by [1], not at all angry, and [5], very angry), and how much they would blame the other person (or persons) (anchored by [1], not at all, and [5], very much). Finally, the participant is asked to write down how she/he would respond to the situation, which is later coded by 2 independent raters to compute an "aggression index."

Social Function Measures (Secondary outcomes) The Specific Levels of Functioning Scale is a 30-item questionnaire that has recently been found to be an excellent measure of social and general real-world functioning. The questionnaire has 2 social functioning subsections (Interpersonal Relationships, Social Acceptability) and 2 community living skills subsections (Activities, Work Skills). One version is completed by the subject and another is completed by an informant, who will meet the following criteria: a) does not have a psychotic disorder, b) is literate, c) has known the subject for at least 1 year, and d) spends time with the subject on a regular basis (e.g., case worker, clinician, family member, caretaker). After giving informed consent, these criteria will be reviewed with each prospective informant. Informants will be compensated for each completed questionnaire. The informant questionnaire asks how well she/he knows the affected participant. Each item is rated on a 5-point Likert scale with anchors describing the frequency of the behavior and/or the patient's level of independence. To informants understand each item on the SLOF, this instrument will be administered by a member of the research team to the informant either in person or, if more convenient, over the phone.

The Social Competence test consists of two 90-second role-plays. The first role-play is an unstructured conversation in which the research confederate plays the role of a new neighbor with whom the subject is instructed to strike up a conversation. In the second role-play, the research confederate plays an upset friend who the subject is instructed to attempt to console. The role plays are recorded and later scored for conversational skills (e.g. overall social skills; affect; speech content, etc) and ability to perceive distress in others (e.g., emotional empathy; cognitive empathy). We have used similar role plays in the past.

The Cyberball Task is a computerized ball tossing game that investigates the effects of being favored and/or ostracized on four fundamental needs; belonging, control, self-esteem, and meaningful existence.

The Interpersonal Perception Task (IPT-15) is a video task that measures non-verbal perception. It consists of a video of 15 brief scenes (28-122 seconds) with are paired with a question with two or three possible answers, allowing the subject to "decode" something important about the people in the scenes.

Empathy and Motivation Measures (Secondary outcomes) The Interpersonal Reactivity Index of empathy is a self-report measure of cognitive and affective empathy. The IRI consists of 28 items where participants rate how well each item describes them using a five point scale. The 28 items yield four subscales: perspective taking (PT), empathic concern (EC), fantasy (F), and personal distress (PD). The PT subscale measures the tendency to take another's point of view (e.g., "I sometimes try to understand my friends better by imagining how things look from their perspective."). The EC subscale measures feelings of sympathy and concern for others (e.g., "I often have tender, concerned feelings for people less fortunate than me."). The F subscale measures the ability to imagine oneself in the role of a fictitious character in books (e.g., "When I am reading an interesting story or novel, I imagine how I would feel if the events in the story were happening to me."). The PD subscale measures personal feelings of anxiety and unease in interpersonal settings (e.g., "Being in a tense emotional situation scares me."). The IRI has been used previously to assess self-reported empathy in individuals with schizophrenia.

Non-social cognitive Measures (Secondary outcome) The Repeatable Battery for the Assessment of Neuropsychological Status will be administered to measure cognitive abilities such as: immediate memory, delayed memory, visual-spatial, language and attention. The assessment takes about 20-25 minutes to complete and will be administered by a trained research assistant. The RBANS will allow us to determine the relationship between neurocognitive abilities and social cognitive abilities, particularly in regards to accuracy in theory of mind testing and emotion perception.

Psychiatric Measures (Secondary outcomes) The Positive and Negative Symptoms Scale is a 30-item scale on which an interviewer rates the subject for severity of positive and negative psychotic symptoms, and general and symptoms after asking a standard series of questions. Items are rated on a scale of 1 (absent) to 7 (severe), and yield five scaled scores: positive symptoms, negative symptoms, dysphoric mood, activation, and autistic preoccupation.

The Green Paranoia Thought Scale consists of two 16-item scales to assess ideas of social reference and persecution.

The Clinical Global Impressions (CGI) Severity Scale is a widely used scale in schizophrenia research for repeated evaluations of global psychopathology. The CGI-S is a single Likert scale rating severity of psychopathology at the time of rating on a scale of 1 (normal, not ill) to 7 (very severely ill). Patients are assessed on the basis of the rater's total clinical experience.

The Calgary Depression Rating Scale is an interviewer-rated measure of depression for individuals with schizophrenia.

The Liebowitz Social Anxiety Scale is a questionnaire that lists 24 social situations on which the subject rates (0-3) how much fear/anxiety he/she would experience and how much he/she would avoid each situation (0-3).

Other Measures Food Cravings and Night Eating Questionnaires. Atypical antipsychotic medications, (which most subjects will be taking), increase appetite and may contribute to weight gain. Oxytocin is known to affect food intake in animals. Therefore, we are including these measures that have been used in previous studies of weight gain/appetite change in patients taking atypical antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yrs of age;
* currently meeting DSM-IV criteria for schizophrenia or schizoaffective disorder with onset occurring > 1 year prior to enrollment in the study;
* score of <24 on the Reading the Mind in the Eyes Test ("Eyes Test", Baron-Cohen, et al 2001), which represents 0.5 SD below the mean in a large normative sample OR
* get a minimum score of "3" on at least two of the following "social" items on the PANSS ratings: suspiciousness/persecution (ideation), hostility, passive/apathetic social withdrawal, uncooperativeness, active social avoidance,
* stable symptoms as well as being on the same medication and psychosocial therapy regimen for > 1 month.

Exclusion Criteria:

* current or lifetime history of schizoaffective (bipolar type), delusional, other psychotic (shared, substance-induced, due to a medical disorder) disorders, bipolar, cyclothymic, somatoform, dissociative, eating or personality disorders, unipolar major depressive episodes with psychotic features, dementia;
* history of mania or hypomania within the past two years
* substance use or abuse disorder during the past 3 months (except tobacco, caffeine);
* treatment currently or within the past 6 months with high dose sedative-hypnotics, stimulants, chronic glucocorticoids (other medications that are adequately controlling acute or chronic disorders [e.g., hypertension, diabetes, hypo or hyperthyroidism, asthma, allergies, mild infections etc.] are allowed);
* debilitating or inadequately controlled medical conditions (including dialysis, HIV infection without AIDS is not exclusionary);
* major surgery/trauma in the past 4 months;
* pregnancy, childbirth or breast-feeding in the past year;
* significant physical exam, laboratory or EKG abnormalities;
* reading level < 5th grade on the Wide Range Achievement Test (WRAT, Wilkinson 1993);
* inability to read English well enough to complete study questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in social cognition scores from baseline to 6 and 12 week time points | Baseline, Week 6, and Week 12 visits

SECONDARY OUTCOMES:
Change in social functioning measures from baseline to 6 and 12 week time points | Baseline, Week 6, and Week 12 visits
Change in PANSS total and subscale scores from baseline to 6 and 12 week time points. | Baseline, Week 6 and Week 12 visits

CONTACTS AND LOCATIONS:
Overall Officials: Cort A Pedersen, MD, Principal Investigator — University of North Carolina, Chapel Hill; David L Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Kohler CG, Turner TH, Gur RE, Gur RC. Recognition of facial emotions in neuropsychiatric disorders. CNS Spectr. 2004 Apr;9(4):267-74. doi: 10.1017/s1092852900009202. PMID 15048051
- [Background] Brüne M (2003) Social cognition and behaviour in schizophrenia. In Brüne M, Ribbert H, Schiefenhövel W (eds.) The social brain-evolution and pathology. John Wiley & Sons; Chichester, pp. 277-313.
- [Background] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Background] Adolphs R, Tranel D, Damasio AR. The human amygdala in social judgment. Nature. 1998 Jun 4;393(6684):470-4. doi: 10.1038/30982. PMID 9624002
- [Background] Combs DR, Penn DL, Wicher M, Waldheter E. The Ambiguous Intentions Hostility Questionnaire (AIHQ): a new measure for evaluating hostile social-cognitive biases in paranoia. Cogn Neuropsychiatry. 2007 Mar;12(2):128-43. doi: 10.1080/13546800600787854. PMID 17453895
- [Background] Schneider LC, Struening EL. SLOF: a behavioral rating scale for assessing the mentally ill. Soc Work Res Abstr. 1983 Fall;19(3):9-21. doi: 10.1093/swra/19.3.9. PMID 10264257
- [Background] Pinkham AE, Penn DL. Neurocognitive and social cognitive predictors of interpersonal skill in schizophrenia. Psychiatry Res. 2006 Aug 30;143(2-3):167-78. doi: 10.1016/j.psychres.2005.09.005. Epub 2006 Jul 21. PMID 16859754
- [Background] Williams KD, Cheung CK, Choi W. Cyberostracism: effects of being ignored over the Internet. J Pers Soc Psychol. 2000 Nov;79(5):748-62. doi: 10.1037//0022-3514.79.5.748. PMID 11079239
- [Background] Davis, MH (1983) Measuring individual differences in empathy: Evidence for a multidimensional approach. J Personal Soc Psychol 44:113-126.
- [Background] Randolph, C. (1998). Repeatable Battery for the Assessment of Neuropsychological Status Manual. San Antonio, TX: Psychological Corporation.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Green CE, Freeman D, Kuipers E, Bebbington P, Fowler D, Dunn G, Garety PA. Measuring ideas of persecution and social reference: the Green et al. Paranoid Thought Scales (GPTS). Psychol Med. 2008 Jan;38(1):101-11. doi: 10.1017/S0033291707001638. Epub 2007 Oct 1. PMID 17903336
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Liebowitz MR. Social phobia. Mod Probl Pharmacopsychiatry. 1987;22:141-73. doi: 10.1159/000414022. No abstract available. PMID 2885745
- [Derived] Merritt CC, Halverson TF, Elliott T, Jarskog LF, Pedersen CA, Penn DL. Racial disparities and predictors of functioning in schizophrenia. Am J Orthopsychiatry. 2023;93(3):177-187. doi: 10.1037/ort0000661. Epub 2023 Mar 16. PMID 36931838